CLINICAL TRIAL: NCT03612479
Title: Response of the Gut Microbiome and Circulating Metabolome to Diet Intervention in Young Children: Ancillary Study to the Keeping Ideal Cardiovascular Health Family Intervention Trial (KIDFIT)
Brief Title: Response of the Gut Microbiome and Circulating Metabolome to Diet in Children: Ancillary Study to KIDFIT (NCT03405246)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: American Heart Association (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Amanda Marma, Assistant Professor in Pediatrics-Cardiology and Preventive Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00207041
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Gastrointestinal Microbiome; Metabolome; Pediatric Obesity; Dietary Approaches to Stop Hypertension
MeSH Terms: conditions — Pediatric Obesity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KIDFIT Healthy (Experimental)
  Interventions: Behavioral: KIDFIT Healthy
- KIDFIT Safe (Active Comparator)
  Interventions: Behavioral: KIDFIT Safe

INTERVENTIONS:
Behavioral: KIDFIT Healthy — The KIDFIT Healthy intervention promotes the DASH diet, physical activity, limited screen time, and adequate sleep, through a combination of traditional in-person and electronic participant contacts. See NCT03405246 for details.
  Other Names: Intervention Group
  Arms: KIDFIT Healthy
Behavioral: KIDFIT Safe — The KIDFIT Safe active control provides electronic material about safe home environments and activities (e.g., sun screen, choking hazards, pet safety) for children. See NCT03405246 for details.
  Other Names: Control Group
  Arms: KIDFIT Safe

SUMMARY:
This is an ancillary study to KIDFIT (NCT03405246). KIDFIT tests whether preschool-age children, born to overweight or obese mothers, respond to a healthy DASH diet intervention with better cardiovascular health.

This ancillary study to KIDFIT investigates how the children's gut microbiomes (bacteria in the intestines) and blood metabolomes (small molecules in the blood) are affected by the DASH diet intervention, and how the microbiome and metabolome relate to the children's cardiovascular health over time. The investigators hypothesize that (1) the DASH diet will modify the gut microbiome and blood metabolome, (2) the gut microbiome and blood metabolome will be related to each other, and (3) the microbiome and metabolome will be associated with the children's cardiovascular health profiles (things like weight, body fat, blood pressure, and cholesterol).

DETAILED DESCRIPTION:
The majority of deaths from cardiovascular disease (CVD) in US adults ages 25-54 years are associated with suboptimal diet. While diet is an important target of CVD prevention efforts in adults, intervention on the childhood diet may be more effective. Animal data suggest that early-life diet has the unique potential to modulate biological systems and durably program a child's biology for long-term health or disease. The objective of this study is to define the molecular effects of a dietary pattern intervention on the gut microbiome and circulating metabolome in young children. This objective will be attained through an ancillary study to KIDFIT, a clinical trial that tests the effects of a 12-month Dietary Approaches to Stop Hypertension (DASH) diet intervention on adiposity and other cardiovascular health (CVH) metrics (e.g., blood pressure, lipids) in 3- to 5-year old children. Using additional participant samples, deep phenotyping and advanced bioinformatics, the ancillary study will address three specific aims. First, it will test the effect of the DASH diet intervention on the gut microbiome, including abundances of microbial taxa, communities, and metabolism-related genes and transcripts. Second, it will define the associations of diet and the gut microbiome with the circulating metabolome. Using targeted and nontargeted metabolomics approaches, blood metabolites, metabolite networks, and metabolic pathways will be evaluated. Finally, in an exploratory fashion, it will probe pathways linking the diet intervention with subsequent adiposity and CVH metrics, through the gut microbiome and serum metabolome. The expected outcome is a preliminary model of how the DASH diet alters the gut microbiome and circulating metabolome in young children, and how these alterations relate to short-term CVH outcomes.

ELIGIBILITY:
Inclusion Criteria:

- participating in KIDFIT (NCT03405246)

Exclusion Criteria:

- none

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Gut microbiome | changes from baseline to 12 months
  abundances of gut microbial taxa, communities, and metabolic pathways activity
Blood metabolome | changes from baseline to 12 months
  abundances of blood metabolites, metabolic networks, and metabolic pathways activity

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Marma Perak, MD MS, Principal Investigator — Northwestern University Feinberg School of Medicine and Ann & Robert H. Lurie Children's Hospital of Chicago
Locations (1):
- Northwestern University Department of Preventive Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH policy to share genomic data from supported studies, raw and processed data from microbiomes, metabolomes, and relevant associated data will be submitted to public data repositories.